CLINICAL TRIAL: NCT02984930
Title: Effect of Proton Pump Inhibitor and Mosapride on Acid Pocket in Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyojin Park, Department of Internal Medicine, Gangnam Severance Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2016-0071
Record Dates: First submitted 2016-08-23; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-08

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole; mosapride; Gastroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPI + mosapride group (Experimental): After diagnosis(GERD), patient of this group will be taken proton pump inhibitor (40mg) plus mosapride for 4weeks. After then, patient of this group will be undergo upper endoscopy and scintigraphy.
  Interventions: Drug: Administration of study drug (esomeprazole, mosapride); Procedure: upper endoscopy, scintigraphy
- PPI + placebo group (Placebo Comparator): After diagnosis(GERD), patient of this group will be taken proton pump inhibitor (40mg) plus placebo drug of mosapride for 4weeks. After then, patient of this group will be undergo upper endoscopy and scintigraphy.
  Interventions: Drug: Administration of study drug (esomeprazole, placebo tablet); Procedure: upper endoscopy, scintigraphy

INTERVENTIONS:
Drug: Administration of study drug (esomeprazole, mosapride) — Esomeprazole(Hanxium®) 40 mg once daily and mosapride (Gasmotin®) 5 mg t.i.d for 4 weeks.
  Arms: PPI + mosapride group
Drug: Administration of study drug (esomeprazole, placebo tablet) — Esomeprazole(Hanxium®) 40 mg once daily and placebo tablets that are identical to mosapride tablets t.i.d (3 times a day) for 4 weeks.
  Arms: PPI + placebo group
Procedure: upper endoscopy, scintigraphy — After medication(4weeks), subjects will be undergo upper endoscopy and scintigraphy.

SUMMARY:
The gastric acid pocket is believed to be the reservoir from which acid reflux events originate. The risk for acidic reflux is mainly determined by the position of the gastric acid pocket. Little is known about how changes in position and size of the acid pocket contribute to the therapeutic effect of proton pump inhibitors(PPI) plus mosapride in patients with gastroesophageal reflux disease. Investigators will conduct a prospective randomized, single blind and placebo-controlled clinical trial to evaluate the hypothesis that mosapride affecting gastric motility might reduce gastro-esophageal reflux by changing the acid pocket position and size.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed GERD(gastro-esophageal reflux disease), defined by the presence of oesophagitis obtained during a previous upper endoscopy or typical GERD symptoms(heartburn, acid reflux).

Exclusion Criteria:

* who had organic gastrointestinal disease including inflammatory bowel disease, cancer and ulcer
* who took drugs which could affect evaluation of the treatment; other PPIs, H2RAs(H2 receptor antagonists), prokinetics,mucosal protective agents, antacids, cholinergic and anticholinergic agents, and antidepressants for at least 4 weeks prior to study start
* who had severe systemic diseases including hepatic and nephrotic disease
* who had previous gastrectomy history
* who was in state of pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Size(cm2) of the acid pocket between PPI+placebo group and PPI+mosapride group | After 4weeks of drug treatment(PPI+placebo vs. PPI + mosapride)
  The size of the acid pocket will be determined by drawing an area of interest over the acid pocket in the proximal stomach in images(scintigraphy) taken at 10-minute intervals.
Location(cm) of the acid pocket between PPI+placebo group and PPI+mosapride group | After 4weeks of drug treatment(PPI+placebo vs. PPI + mosapride)
  Measurements of the distances between the acid pocket and the diaphragm will be make through a straight line in a planar posterior view of the stomach in images(scintigraphy)

SECONDARY OUTCOMES:
Improvement of reflux symptom | After 4weeks of drug treatment(PPI+placebo vs. PPI + mosapride)
  Using RDQ(Reflux Disease Questionnaire)

IPD SHARING:
Plan to Share IPD: No